CLINICAL TRIAL: NCT07199881
Title: Assessment of Respiratory Drive and Inspiratory Effort Across Pressure Support Levels in Patients After Major Abdominal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Siriraj Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PSV-SICU_SIRIRAJ
Record Dates: First submitted 2025-09-10; First posted 2025-09-30 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Inspiratory Effort; Mechanical Ventilation; Major Abdominal Surgeries
Keywords: Pressure support ventilation; respiratory drive; inspiratory effort; mechanical ventilation; Major Abdominal Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Cohort (Postoperative SICU patients on PSV >48h) (Experimental): Adult patients admitted to the surgical ICU after major abdominal surgery who remain on pressure support ventilation (PSV) for more than 48 hours. Each participant will undergo a standardized stepwise protocol of PSV adjustment (baseline, -6 cmH₂O, -3 cmH₂O, +3 cmH₂O, +6 cmH₂O, return to baseline). At each step, a 2-minute stabilization is followed by repeated measurements of respiratory drive and inspiratory effort indices (P0.1, Pocc, PMI) and ventilatory parameters.
  Interventions: Procedure: Stepwise PSV adjustment protocol

INTERVENTIONS:
Procedure: Stepwise PSV adjustment protocol — Patients will undergo standardized stepwise PSV changes (baseline, ±3 cmH₂O, ±6 cmH₂O, return to baseline), with 2-minute stabilization and repeated measurements of ventilatory parameters.

SUMMARY:
This physiological observational study will assess respiratory drive and inspiratory effort across varying levels of pressure support ventilation (PSV) in adult surgical ICU (SICU) patients after major abdominal surgery. By using non-invasive bedside indices (airway occlusion pressure at 100 ms after the onset of inspiration [P0.1], maximum negative occlusion pressure [Pocc], and pressure muscle index [PMI]), we aim to quantify how patients adapt to changes in ventilatory support and determine patterns of under- and over-assistance. Findings may inform optimal titration of PSV to reduce complications and improve clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) admitted to the surgical ICU
* Recent major abdominal surgery (intra-peritoneal operation without primary thoracic involvement, including luminal resection and/or resection of a gastrointestinal solid organ) requiring postoperative ICU care
* Receiving invasive mechanical ventilation in pressure support ventilation (PSV) mode at the time of enrollment
* Duration of invasive mechanical ventilation >48 hours
* Clinically stable, with no plan for extubation within 6 hours of study enrollment, defined by all of the following: Respiratory rate <35 breaths/min, SpO₂ ≥90%, Heart rate <140 bpm, No visible accessory muscle use, Hemodynamically stable without escalation of vasopressor support during the past hour, Able to tolerate short-term adjustments in PSV level as per protocol

Exclusion Criteria:

* Known neuromuscular disease affecting respiratory muscle function
* Hemodynamic instability requiring escalation of vasopressor support
* Severe hypoxemic respiratory failure requiring Positive End-Expiratory Pressure (PEEP) >10 cmH₂O or FiO₂ >60%
* Deep sedation (Richmond Agitation-Sedation Scale [RASS] score < -3) or ongoing neuromuscular blockade
* History of chronic obstructive pulmonary disease (COPD) or other obstructive lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Respiratory drive and inspiratory effort across pressure support levels | Baseline and during protocol sessions, up to 3 days after enrollment
  Respiratory drive and inspiratory effort will be assessed using airway occlusion pressure at 0.1 seconds (P0.1), maximum negative inspiratory occlusion pressure (Pocc), and the pressure muscle index (PMI). These indices are measured non-invasively via ventilator maneuvers during standardized stepwise adjustments of pressure support ventilation (baseline, ±3 cmH₂O, ±6 cmH₂O, return to baseline). The mean of three repeated measurements at each step will be analyzed.

SECONDARY OUTCOMES:
Incidence of ventilatory response patterns during PSV | Baseline and during protocol sessions, up to 3 days after enrollment
  Ventilatory response patterns will be categorized as quasi-passive or active based on physiological criteria derived from changes in tidal volume, plateau pressure, and PMI during stepwise PSV adjustments. Patterns will be determined from individual response trends.
Duration of mechanical ventilation after protocol | Within 48 hours after extubation
  Time from completion of the PSV protocol until successful extubation, measured in hours. Reintubation within 48 hours will be recorded separately.
Reintubation or non-invasive ventilation use | 48 hours after extubation
  Proportion of patients requiring reintubation or initiation of non-invasive ventilation within 48 hours after extubation following study participation.
ICU length of stay | Through ICU stay, an average of 7-21 days
  Total number of days from ICU admission to ICU discharge.
Hospital discharge disposition | Through hospital stay, an average of 14-60 days
  Patient's status at hospital discharge (alive vs. deceased; home vs. rehabilitation vs. long-term care).

CONTACTS AND LOCATIONS:
Overall Officials: Nuanprae Kitisin, Principal Investigator — Department of Anesthesiology, Faculty of Medicine, Siriraj Hospital, Mahidol University
Locations (1):
- Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok, Bangkoknoi, Thailand

IPD SHARING:
Plan to Share IPD: No
This is a single-center physiological observational study with a modest sample size. No plan to share individual participant data outside the study team. Summary data will be available in publications

REFERENCES:
- [Result] He Q, Lai Z, Peng S, Lin S, Mo G, Zhao X, Wang Z. Postoperative pulmonary complications after major abdominal surgery in elderly patients and its association with patient-controlled analgesia. BMC Geriatr. 2024 Sep 10;24(1):751. doi: 10.1186/s12877-024-05337-y. PMID 39256677
- [Result] Miskovic A, Lumb AB. Postoperative pulmonary complications. Br J Anaesth. 2017 Mar 1;118(3):317-334. doi: 10.1093/bja/aex002. PMID 28186222
- [Result] Courtney A, Clymo J, Dorudi Y, Moonesinghe SR, Dorudi S. Scoping review: The terminology used to describe major abdominal surgical procedures. World J Surg. 2024 Mar;48(3):574-584. doi: 10.1002/wjs.12084. Epub 2024 Feb 11. PMID 38342951
- [Result] Docci M, Foti G, Brochard L, Bellani G. Pressure support, patient effort and tidal volume: a conceptual model for a non linear interaction. Crit Care. 2024 Nov 6;28(1):358. doi: 10.1186/s13054-024-05144-2. PMID 39506755
- [Result] Al-Bassam W, Parikh T, Neto AS, Idrees Y, Kubicki MA, Hodgson CL, Subramaniam A, Reddy MP, Gullapalli N, Michel C, Matthewman MC, Naughton J, Pereira J, Shehabi Y, Bellomo R. Pressure support ventilation in intensive care patients receiving prolonged invasive ventilation. Crit Care Resusc. 2023 Oct 18;23(4):394-402. doi: 10.51893/2021.4.OA4. eCollection 2021 Dec 6. PMID 38046681
- [Result] van Oosten JP, Akoumianaki E, Jonkman AH. Monitoring respiratory muscles effort during mechanical ventilation. Curr Opin Crit Care. 2025 Feb 1;31(1):12-20. doi: 10.1097/MCC.0000000000001229. Epub 2024 Nov 14. PMID 39560150

DOCUMENTS (1):
  • Study Protocol (2025-09-17): https://cdn.clinicaltrials.gov/large-docs/81/NCT07199881/Prot_000.pdf